CLINICAL TRIAL: NCT03105245
Title: Understanding How Anaesthesia Affects ECT Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Wesley Mission (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HREC16952
Record Dates: First submitted 2017-02-27; First posted 2017-04-07 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: electroconvulsive therapy; anaesthesia
MeSH Terms: conditions — Depression | interventions — Electroconvulsive Therapy; Anesthetics; Thiopental

STUDY DESIGN:
Intervention Model Description: Each participant will receive all four treatment conditions in randomly allocated sequence during their ECT course. That is, participants will receive either short or long anaesthetic-ECT stimulus time interval treatments, and normal or hyperventilation treatments - this results in four possible combinations, which individual participants will cycle through in random order during their ECT course (e.g. short-hyperventilation, long-normal ventilation, short-normal ventilation, long-hyperventilation).
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and the outcome assessor (analysing EEGs) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Short time interval + Normal ventilation (Active Comparator)
  Interventions: Other: Electroconvulsive Therapy (ECT) time interval + Anaesthetic (Thiopentone)
- Short time interval + Hyperventilation (Active Comparator)
  Interventions: Other: Electroconvulsive Therapy (ECT) time interval + Anaesthetic (Thiopentone)
- Long time interval + Normal ventilation (Active Comparator)
  Interventions: Other: Electroconvulsive Therapy (ECT) time interval + Anaesthetic (Thiopentone)
- Long time interval + Hyperventilation (Active Comparator)
  Interventions: Other: Electroconvulsive Therapy (ECT) time interval + Anaesthetic (Thiopentone)

INTERVENTIONS:
Other: Electroconvulsive Therapy (ECT) time interval + Anaesthetic (Thiopentone) — The intervention in this study is the time interval between anaesthetic administration and ECT stimulus

SUMMARY:
This study will examine how anaesthetic technique affects ECT outcomes. Specifically, the investigators will examine how: 1) the time interval between anaesthetic and ECT stimulus, and 2) the ventilation rate before ECT stimulus, impacts on the quality of the EEG (this is a recording of brain activity during ECT and is used to judge the quality of a seizure and to guide individual patient dosing).

DETAILED DESCRIPTION:
This study aims to examine how the time interval between administration of anaesthetic agent and ECT stimulus delivery impacts upon measures of EEG quality (seizure quality).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with a course of ECT

Exclusion Criteria:

* Use of non-standard anaesthetic agents in ECT (e.g. ketamine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
EEG Seizure Quality Rating using the EEG Seizure Quality Rating Sheet utilised by MacPherson et al | Outcome measures will be collected immediately after each ECT treatment from the first treatment until the end of the ECT course, an estimated total of four to six weeks for most participants
  EEG quality will be rated manually for each ECT treatment undertaken by a participant until the conclusion of their ECT course. This rating will be done using the EEG Seizure Quality Rating Sheet utilised by MacPherson et al - low dose lignocaine added to propofol does not attenuate the response to electroconvulsive therapy; Journal of Affective Disorders, 2010; 126: 330-333

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, Principal Investigator — The University of New South Wales
Locations (1):
- Wesley Hospital Kogarah, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No